CLINICAL TRIAL: NCT03159039
Title: Study of Clinical Repercussions of Conventional Respiratory Physiotherapy Versus Prolonged Slow Expiration in Preterms Under Mechanical Ventilation
Brief Title: Repercussions of Respiratory Physiotherapy in Preterm Infants Under Mechanical Ventilation
Acronym: preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Viviani Barnabe, Dr, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: preterm physiotherapy
Record Dates: First submitted 2017-04-06; First posted 2017-05-18 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Drainage, Postural

STUDY DESIGN:
Intervention Model Description: Patients will randomized in 2 groups: group CCP (conventional chest physiotherapy techniques) (n=22) , the technique will made during 5 minutes in each side and after that, endotraqueal aspiration will performed.or group PSE (prolonged slow exhalation technique) (n=21), the technique will made during 10 minutes, 2 times a day.At the end, endotraqueal aspiration will perfomed.
  During the protocol the parameters will recorder: respiratory rate, heart rate and peripheral oxygen saturation, exhaled tidal volume, number of days under mechanical ventilation and number of fail times in extubation. In 5 diferent moments.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy (PT) (Experimental): Postural drainage + manual vibration
  Interventions: Other: Conventional Physiotherapy
- Prolonged slow exhalation technique (Active Comparator): Prolonged exhalation + Conventional PT
  Interventions: Other: Prolonged slow exhalation technique

INTERVENTIONS:
Other: Conventional Physiotherapy
  Other Names: Postural drainage
  Arms: Conventional Physiotherapy (PT)
Other: Prolonged slow exhalation technique — Postural drainage associated with manual vibration and a mild pressure in the end of expiratory phase
  Arms: Prolonged slow exhalation technique

SUMMARY:
Respiratory diseases are a major morbidity and mortality causes of neonatal requiring mechanical ventilation, especially in newborn preterm infants (PN), thus respiratory therapy becomes increasingly necessary in order to minimize the effects of complications and improve respiratory functions, increasing mucociliary transport with techniques that consist of manual maneuvers to bronchial hygiene, such as vibro associated with postural drainage and prolonged slow exhalation. Objective: To compare and analyze the effects of convensional physiotherapy (CP) versus prolonged slow exhalation (PSE) in heart rate (HR), and respiratory rate (RR), O2 saturation (SpO2) and Tidal Volume (TV), time permanence of mechanical ventilation (TMV) and number of extubation failure (EF) in premature infants on mechanical ventilation (MV). Methods: Randomized clinical trial conducted in the neonatal intensive care unit of the General Hospital Itapecerica da Serra Seconci OSS SP, comparing two physical therapy techniques applied to preterm infants on mechanical ventilation.

DETAILED DESCRIPTION:
Neonates patients admitted at unit of Intensive Care of Geral Hospital of Itapecerica da Serra (São Paulo-Brazil) will recruited to this study. Based on World Health Organization (WHO), the neonates preterm are those who present gestational age (GA) <35 weeks (gestational age was calculated based on the date of last menstruation). Inclusion criteria: neonates born at GA<35 weeks, under mechanical ventilation (interplus 5 -Intermédica® or servo i (Maquet, Solvan, Sweden) for the first 7 days of life, hemodynamically stable; birth weight ≤1.500 gram; per cent change inspired oxygen received (FiO2) ≤ 0.6; Inspiratory pressure ≥ 25 cmH2O; medical prescription of chest physiotherapy. Exclusion criteria: congenital malformation graves; genetic syndromes and situations, pulmonary hypertension, peri-intraventricular hemorrhage and coagulopathies.

All patients will receive chest physiotherapy when it is necessary and all of them will monitored until dischange.

After performed all included criteria, patients will randomized in 2 groups: group CCP (patients submitted to conventional chest physiotherapy techniques) or group PSE (patients submitted to prolonged slow exhalation technique).

After that, for both group, physiotherapist take note of gestacional age, gender, bith weight (gram), Apgar score (1º; 5º and 10º minute), type of delivery, medical diagnosis, mechanical ventilation parameters, medications. Then, lung auscultation, breathing pattern, pulse oximetry and radiological chest pattern of all patients will evaluated by the same physiotherapist.

CCP group (n=22): patients will submitted to a postural drainage associated with manual vibration. They will positionated with left or right of ribcage to up and then physiotherapist made a manual vibratory movements associated with a mild compression in ribcage at the end of expiratory phase. The technique was made during 5 minutes in each side. After that, endotraqueal aspiration will performed.

PSE group (n=21): patients will carefully positionated with head up (30º) and then physiotherapist put one hand around ribcage area e another in abdominal area then he made a mild pressure in both areas at the same time in the end of expiratory phase of patient until residual volume keeping the pressure for 2 seconds. This technique will made during 10 minutes.At the end, endotraqueal aspiration will perfomed.

Both techniques will realized with the same physiotherapist, 2 times a day (morning and afternoon) during 10 minutes and all data were recorded during the 2 first days of physiotherapy assistance.

During the protocol, the follow data will recorded: respiratory rate (digital timer C4539-Brady, Brazil), heart rate and peripheral oxygen saturation (multiparameter monitor DX 2010 -Dixtal Biomédica, Brazil), exhaled tidal volume (internal sensor ventilation mechanical), number of days under mechanical ventilation and number of fail times in extubation. These parameters will recorded in 5 diferent moments: T0 (before beginning of physiotherapy);T1 (immediately after physiotherapy technique); T2 (immediately after cannula aspiration); T3 (after 5 minutes of all procedures); T4 (20 minutes after all procedures).

ELIGIBILITY:
Inclusion Criteria:

• Preterms born at gestational age <35 weeks under mechanical ventilation

Exclusion Criteria:

* congenital malformation graves;
* genetic syndromes,
* pulmonary hypertension,
* peri-intraventricular haemorrhage and coagulopathies.

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — gestational age (GA) <35 weeks
Enrollment: 43 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Tidal volume | 10 minutes twice a day
  Measured by the mechanical ventilator

SECONDARY OUTCOMES:
Respiratory rate | 10 minutes twice a day
  Measured by the mechanical ventilator

OTHER OUTCOMES:
Peripheral oxygen saturation | 10 minutes twice a day
  Measured by the oxymeter
Heart rate | 10 minutes twice a day
  Measured by the oxymeter

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Sraiva-Romanholo, PhD, Study Chair — Universidade Cidade de Sao Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blencowe H, Cousens S, Chou D, et al. Born Too Soon: The global epidemiology of 15 million preterm births. Reproductive Health. 2013;10(Suppl 1):S2. doi:10.1186/1742-4755-10-S1-S2. Beck , Wojdyla LS, Betran AP, Merialdi M, Requejo JH, Rubens C, et al. The worldwide incidence of preterm birth: a systematic review of maternal mortality and morbidity. Bull World Health Organ. 2010; 88:31-8. Koivisto M, Marttila R, Kurkinen-Raty M, Saarela T, Pokela ML, Jouppila P, et al. Changing incidence and outcome of infants with respiratory distress syndrome in the 1990s: a population-based survey. Acta Paediatr. 2004; 93: 177-184. Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet .2008;371:75-84. Kamath BD, MacGuire ER, McClure EM, Goldenberg RL, Jobe AH. Neonatal Mortality From Respiratory Distress Syndrome: Lessons for Low-Resource Countries. Pediatrics.2011;127:1139-1146. doi: 9.1542/peds.2010-3212 10. Sweet, David G., et al.